CLINICAL TRIAL: NCT05061238
Title: Impact Of Muscle Vibration On Gait Control
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-0620; NCI-2021-09935 (Other: NCI-CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2021-09-16; First posted 2021-09-29 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Muscle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Vibrating Device (Other): you will be asked to walk up and down a hallway 5 times with the vibrating device strapped to different parts of your leg.
  Interventions: Device: Vibrating Device

INTERVENTIONS:
Device: Vibrating Device — The vibrating device strapped to different parts of your leg. The device will be secured to your leg with a Velcro strap.

SUMMARY:
This is a single-site interventional open label pilot study of a non-significant risk medical device on patients with defined peripheral neuropathy secondary to chemotherapy (N=10). Patients who have received chemotherapy and have evidence of neuropathy will be seen at MD Anderson. Their severity of neuropathy will be documented and assessed by physical therapy, occupational therapy and based on self-reported activities of daily living (ADL) impairment.

DETAILED DESCRIPTION:
Primary Objective:

To assess the effect of a vibrating device applied to selected muscles on the step

Secondary Objectives:

* To summarize the adverse events of different levels from using the vibrator device in oncologic AYA patients visiting the outpatient clinic.
* To summarize the irritation, pain, and sensation of the application of vibration by the AYA patients, as determined by the survey during the application

ELIGIBILITY:
Inclusion Criteria:

* Subjects between the ages of 6 and 39 years.
* Study subjects, or their parent/legal guardian for subjects <18 years, must be able to understand the purpose and risks of the study and to provide signed and dated informed consent and authorization to use confidential health information in accordance with national and local subject privacy regulations.
* History of any type of cancer-
* Diagnosed with peripheral neuropathy-associated gait dysfunction as defined by the treating physician.
* Able (in the Investigators estimation) and willing to comply with all study requirements.
* Subjects must be able to walk; assistance of a walker or similar support apparatus is allowed.
* Patients with ankle foot orthosis (AFOs) are allowed but will need to be removed prior to testing.

Exclusion Criteria:

* Participants with amputations, prosthetics, congenital malformations or any severe lower extremity deformities affecting gait before trials.
* Abnormalities of the lower extremities as determined by the investigator.
* Unstable participants or participants with hypotension (systolic blood pressure <90 and diastolic blood pressure < 60mmHg).
* Any other significant disease or disorder which, in the opinion of the investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Other unspecified reasons that, in the opinion of the Investigator make the subject unsuitable for enrolment
* Pregnant women
* Children <15 years old
* Blind

Ages: 6 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To establish the effect of a vibrating device applied to selected muscles on the step times of adolescent or young adult (AYA). | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: David McCall, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org